CLINICAL TRIAL: NCT02245425
Title: A Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain: A Randomized Controlled Trial
Brief Title: Comparison of Two Thoracic Manipulation Techniques to Improve Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014096
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Neck Pain
Keywords: Neck pain; Thoracic spine manipulation; Range of Motion; Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supine Thoracic Spine Manipulation (Active Comparator): Supine (lying face-up on the treatment table) thoracic spine thrust manipulation will be given 2 times at 3 treatment sessions (Weeks 0, 1, and 2)
  Interventions: Other: Supine Thoracic Spine Manipulation
- Prone Thoracic Spine Manipulation (Active Comparator): Prone (lying face down on the treatment table) thoracic spine thrust manipulation will be given 2 times at 3 treatment sessions (Weeks 0, 1, and 2).
  Interventions: Other: Prone Thoracic Spine Manipulation

INTERVENTIONS:
Other: Supine Thoracic Spine Manipulation — Position patient so that small amplitude quick stretch can be applied to the least mobile area of the thoracic spine that is identified during the spinal segmental mobility testing. The thoracic spine thrust manipulation will be applied at an appropriate range of motion as identified by the clinician.
  Arms: Supine Thoracic Spine Manipulation
Other: Prone Thoracic Spine Manipulation — Position patient so that small amplitude quick stretch can be applied to the least mobile area of the thoracic spine that is identified during the spinal segmental mobility testing. The thoracic spine thrust manipulation will be applied at an appropriate range of motion as identified by the clinician.
  Arms: Prone Thoracic Spine Manipulation

SUMMARY:
This study is designed to compare the short-term effects of two different thoracic spine thrust manipulation techniques on neck range-of-motion, pain, and self-reported disability in people with neck pain.

The null hypothesis is that there will be no differences between the two manipulation techniques for short-term effects on neck range-of-motion, pain, and self-reported disability in people with neck pain.

DETAILED DESCRIPTION:
Patients will be involved in the study over a 4 week period. Each participant will be asked to attend 4 sessions, with one week in between each session as follows: Week 0 = baseline assessment and treatment 1; Week 1= treatment 2; Week 2 = treatment 3; and week 4 = follow-up assessment.

Patients who meet the inclusion/exclusion criteria will be randomized to either a supine or prone thoracic spine thrust manipulation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between 22 and 50 years of age
* Primary complaint of neck pain with or without symptoms that spread down into one arm
* Overall rating of neck pain intensity is at least 3/10; the overall rating is the overall average of the participant's rating of current, least, and worst pain experienced over the previous 24 hours on separate numeric pain rating scales where 0 corresponds to "no pain" and 10 corresponds to "worst pain possible".
* Neck Disability Index (NDI) score > 10 points (measure of self-reported disability with a 0 to 50 point scale where higher scores indicate higher levels of disability).
* Proficient in speaking and reading English to complete outcome questionnaires

Exclusion Criteria:

* Neck pain related to a motor vehicle accident or other trauma within the previous 6 weeks
* Neck pain that spreads down into both arms
* Low back pain or thoracic origin of pain
* Nerve root involvement; defined as the presence of two or more neurological findings (e.g. decreased strength, diminished deep tendon reflex, or decreased sensation) at the same nerve root level
* Diagnosis of cervical spine stenosis (narrowing of the central canal that contains the spinal cord)
* History of spinal tumors, spinal infection, cervical spine fracture, or previous neck surgery
* Pending legal action related to current episode of neck pain
* Contraindications to thoracic spine thrust manipulation

  1. serious pathologies or conditions (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, history of prolonged steroid use)
  2. hyperreflexia
  3. unsteadiness during gait
  4. Nystagmus
  5. Loss of visual acuity
  6. Impaired sensation of the face
  7. Altered taste
  8. The presence of pathological reflexes
  9. pregnancy or considering pregnancy

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04-30 (Actual); Study Completion 2015-07-08 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline (Week 0)
  Patient-rated assessment of pain on scale of 0-10
NPRS | Change from Week 0 to Week 1
  Patient-rating of pain on a scale of 0-10
NPRS | Change from Baseline (Week 0) and Follow-up (Week 3) and From Week 1 and Week 3
  Patient-rating of pain on a scale of 0-10
Neck Disability Index (NDI) | Baseline (Week 0)
  10 Question patient-rated outcome measures specific to neck disability
NDI | Change from Baseline (Week 0) to Week 1
  10 Question patient-rated outcome measures specific to neck disability
NDI | Change from Baseline (Week 0) to Follow-up (Week 3) and from Week 1 to Week 3
  10 Question patient-rated outcome measures specific to neck disability
Shortened Version of Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) | Baseline (Week 0)
  11 item patient-rated outcome measure related to disability in the upper extremity with optional work and sport modules.
QuickDASH | Change from Week 0 to Week 1
  11 item patient-rated outcome measure related to disability in the upper extremity with optional work and sport modules.
QuickDASH | Change from Baseline (Week 0) to Follow-up (Week 3) and from Week 1 to Week 3
  11 item patient-rated outcome measure related to disability in the upper extremity with optional work and sport modules.
Neck Range of Motion (ROM) | Baseline (Week 0)
  Cervical rotation and lateral flexion measured with goniometer.
Neck ROM | Change from Baseline (Week 0) to Week 1
  Cervical rotation and lateral flexion measured with goniometer.
Neck ROM | Change from Baseline (Week 0) to Follow-up (Week 3) and between Week 1 and Week 3
  Cervical rotation and lateral flexion measured with goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: John Heick, PT, DPT, Principal Investigator — A.T. Still University
Locations (1):
- A.T. Still University, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No